CLINICAL TRIAL: NCT04060667
Title: Wireless Physiologic Monitoring in Postpartum Women
Acronym: WIMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Adeline A Boatin, Assistant Professor of OB/GYN, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019P000885; K23HD097300-01 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-19 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Maternal Death During Childbirth; Pregnancy Complications
Keywords: vital sign monitoring; maternal near miss; maternal mortality; maternal morbidity; physiologic monitoring; quality of care; inpatient monitoring
MeSH Terms: conditions — Pregnancy Complications; Maternal Death

STUDY DESIGN:
Intervention Model Description: describe time blocks, include description of time allotment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm were monitored for up to 24 hours after an emergency cesarean section using the Current Health wireless physiologic monitoring system, which includes a wearable biosensor that records heart rate, temperature, respiratory rate, oxygen saturation, and movement continuously and transmits data in real-time via a wireless network to the cloud.
  Interventions: Combination Product: Wireless physiologic monitoring
- control (No Intervention): Participants in the control arm had standard of care monitoring, using available tools on the wards (manual heart rate, temperature, and respiratory rate calculations).

INTERVENTIONS:
Combination Product: Wireless physiologic monitoring — The intervention in this study is the use of a wireless monitor to perform physiologic monitoring of women undergoing emergency cesarean delivery for the first 24 hours after completion of the cesarean and send alerts to responding clinicians should vital signs fall out of a pre-specified range.
  Other Names: vital sign abnormality alerts
  Arms: Intervention

SUMMARY:
To estimate the clinical effectiveness of wireless physiologic monitoring of women in the first 24 hours after cesarean delivery at Mbarara Regional Referral Hospital

DETAILED DESCRIPTION:
Women in sub-Saharan Africa have the highest rates of morbidity and mortality during childbirth. Despite significant increases in facility-based childbirth, quality gaps at the facility have limited reductions in maternal deaths. Infrequent monitoring of women around childbirth is a major gap in care that leads to delays in life-saving interventions. Simple increases in staffing will not overcome this gap, thus necessitating new strategies.

This project aims to use a simple wireless monitor to improve the detection of complications immediately after childbirth and allow clinicians to provide life-saving interventions when needed. Using a hybrid clinical effectiveness-implementation approach women delivered by cesarean in Mbarara, Uganda will be recruited to wear a wireless physiologic monitor for 24 hours after delivery and their delivering obstetricians recruited to use the monitoring system, including the receipt of text message alerts should women develop abnormalities in physiologic signs. Rates of morbidity and mortality will be compared with a control group of women delivered by the same obstetricians. Clinical adoption and implementation will be assessed with the RE-AIM implementation framework and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Emergency cesarean delivery at MRRH
* Able to provide consent or have a guardian/attendant present who can consent
* Willing to wear the biosensor for 24 hours
* Willing remain in the postpartum unit for 24 hours

Exclusion Criteria:

* Admitted to ICU directly after delivery
* Allergies or hypersensitivity to device materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3191 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline A Boatin, MD MPH, Principal Investigator — MGH
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boatin AA, Ngonzi J, Wylie BJ, Lugobe HM, Bebell LM, Mugyenyi G, Mohamed S, Martinez K, Musinguzi N, Psaros C, Metlay JP, Haberer JE. Wireless versus routine physiologic monitoring after cesarean delivery to reduce maternal morbidity and mortality in a resource-limited setting: protocol of type 2 hybrid effectiveness-implementation study. BMC Pregnancy Childbirth. 2021 Feb 12;21(1):124. doi: 10.1186/s12884-021-03550-w. PMID 33579213

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a study in which a single health facility was assigned to alternating two-week "intervention" and "control" periods. During the intervention periods, participants were consented, and received the study intervention. During the control periods, participants received standard of care and medical record review only was performed. Consent was waived for participants in the control periods.
Groups:
- Intervention: Wireless Physiologic Monitoring
- Control: Standard of Care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1552 | 1639
Completed | 1477 | 1629
Not Completed | 75 | 10
Not completed — Lost to Follow-up | 75 | 10

BASELINE CHARACTERISTICS:
Groups:
- Control: Standard of Care monitoring
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1552 | 1629 | 3181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1552 | 1629 | 3181
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (5.4) | 26.6 (5.8) | 26.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1552 | 1629 | 3181
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Parity [Mean (Standard Deviation); unit: number of pregnancies] | 2.2 (1.6) | 2.2 (1.5) | 2.2 (1.5)
Gestational Age [Mean (Standard Deviation); unit: completed weeks of gestation] — Population: Missing data
  completed weeks of gestation
    number analyzed (Participants) | 1546 | 1629 | 3175
    (all) | 39.1 (2.5) | 39.2 (2.5) | 39.1 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Severe Maternal Outcome
Description: The primary effectiveness outcome was a composite measure of severe maternal morbidity (SMM) measured from enrollment until hospital discharge This composite measure is adapted from World Health Organization (WHO) near-miss morbidity criteria, as well as other severe maternal outcomes, including hysterectomy, cardiac arrest, prolonged unconsciousness, stroke, dialysis, intensive care admission, and death.
Time Frame: From completion of the cesarean delivery until hospital discharge from the procedure, an average of 3 days
Population: Analysis was restricted to participants consenting for participation (intervention group) or with completed medical record review (control group)
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1552 | 1639
participants | 25 | 25

ADVERSE EVENTS:
Time Frame: Until hospital discharge, an average of 3 days
Description: Our primary outcome measure was severe maternal outcome; the outcomes collected as part of this composite outcome include: blood transfusion, hysterectomy, cardiac arrest, prolonged unconsciousness, stroke, dialysis, intensive care admission, and death
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 3/1552 | 1/1629
Serious Adverse Events (participants affected / at risk) | 6/1552 | 12/1629
Other Adverse Events (participants affected / at risk) | 0/1552 | 0/1629
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1552) | Control (N=1629)
Hysterectomy (Reproductive system and breast disorders) | 3 (3) | 6 (6) — Removal of the uterus
Re-operation (Surgical and medical procedures) | 1 (1) | 2 (2) — Need for re-operation after the initial surgery (cesarean delivery)
ICU admission (Surgical and medical procedures) | 2 (2) | 3 (3) — admission to the intensive care unit
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — need for cardiopulmonary resuscitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT04060667/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04060667/SAP_001.pdf